CLINICAL TRIAL: NCT04841395
Title: Morningness Chronotype is Associated With Premature Ejaculation
Brief Title: Chronotype and Premature Ejaculation
Status: Completed | Type: Observational
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Sinay Önen, Associate Professor, Bursa Yuksek Ihtisas Training and Research Hospital
Other Study IDs: 2011-KAEK-25 2019/04-18
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PE: Premature ejaculation group
  Interventions: Diagnostic Test: Intravaginal ejaculatory latency time (IELT), Arabic Index of Premature Ejaculation (AIPE), Morningness-Eveningness Questionnaire (MEQ)
- CG: Control group (Healthy subjects)
  Interventions: Diagnostic Test: Intravaginal ejaculatory latency time (IELT), Arabic Index of Premature Ejaculation (AIPE), Morningness-Eveningness Questionnaire (MEQ)

INTERVENTIONS:
Diagnostic Test: Intravaginal ejaculatory latency time (IELT), Arabic Index of Premature Ejaculation (AIPE), Morningness-Eveningness Questionnaire (MEQ) — Self-estimated intravaginal ejaculatory latency time IELT is defined as the time between the onset of vaginal intromission and the onset of intravaginal ejaculation. In the present research, self-estimated IELT duration was obtained as a result of interviews with the participants. Moreover, Arabic Index of Premature Ejaculation (AIPE), International Index of Erectile Function (IIEF-5), Pittsburgh Sleep Quality Index (PSQI) and Morningness-Eveningness Questionnaire (MEQ) were administered to all participants.

SUMMARY:
Chronotype (or circadian preference) has previously been shown to be associated with sexual attitudes and behaviors and is an important factor affecting sexual satisfaction. The fact that some neurobiological variables, which are thought to have a role in ejaculation physiology, are also effective in the processes of sleep and the regulation of circadian rhythm, and evidence supporting the relationship between circadian preferences and sexual desire and sexual behavior; suggests that ejaculation disorders may be related to circadian preference. The aim of the present study was to investigate the relationship between intravaginal ejaculatory latency time (IELT), severity of disease and chronotype in lifelong PE.

DETAILED DESCRIPTION:
After being informed about the study, all patients who gave written informed consent were questioned and diagnosed as lifelong PE according to the definition of International Society of sexual medicine (ISSM) by an experienced urologist. Since erctile dysfunction (ED) may accompany PE, the presence of ED symptoms was evaluated by the International Index of Erectile Function (IIEF-5), and those with IIEF-5 score <22 were excluded from the study. Age- and sex-matched control cases without lifelong PE were selected randomly among cases attending the hospital for a checkup procedure. A total of 114 patients with PE and 103 control subjects with similar sociodemographic characteristics were included in the study. A detailed medical and sexual history was taken, which included self-estimated intravaginal ejaculatory latency time (IELT), by an experienced sexual therapist. Moreover, Arabic Index of Premature Ejaculation (AIPE), Pittsburgh Sleep Quality Index (PSQI) and Morningness-Eveningness Questionnaire (MEQ) were administered to all participants.

ELIGIBILITY:
Inclusion Criteria:

* male between the ages of 18-50 years,
* being sexually active, and in a stable relationship with a single partner for the last 6 months
* meeting diagnostic criteria of Premature ejaculation according to ISSM.

Exclusion Criteria:

* having a history of neurological and/or psychiatric disorders, any malignancies, sexual dysfunction other than PE, chronic systemic disease, or if they were taking alpha-blockers, phosphodiesterase type-5 inhibitors, 5-alpha reductase inhibitors, anticholinergics, antipsychotics, or antidepressants.
* presence of obesity (body mass index (BMI)> 30)
* presence of Erectile Dysfunction (IIEF-5 score <22)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self representation of male gender, sexually active, and in a stable relationship with a single partner for the last 6 months.
Study Population: Males who presented at the outpatient clinic of Urology with the self-reported complaint of lifelong premature ejaculation
Sampling Method: Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
MEQ scores | Baseline
  MEQ is a measurement tool developed to measure the morning and evening sleep cycle associated with circadian rhythm (Horne & Östberg, 1976). It consists of 19 self-reported likert-type items and has a rating range from 16 to 86. Higher scores in the MEQ refer to morningness chronotype, and lower scores refer to eveningness chronotype. In the Turkish adaptation study of MEQ, three different categories of circadian rhythm were defined as; 59-86 points "morningness type", 42-58 points "intermediate type", 16-41 points "eveningness type"

CONTACTS AND LOCATIONS:
Overall Officials: Efe Önen, M.D., Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jankowski KS, Diaz-Morales JF, Randler C. Chronotype, gender, and time for sex. Chronobiol Int. 2014 Oct;31(8):911-6. doi: 10.3109/07420528.2014.925470. Epub 2014 Jun 13. PMID 24927370
- [Background] Jocz P, Stolarski M, Jankowski KS. Similarity in Chronotype and Preferred Time for Sex and Its Role in Relationship Quality and Sexual Satisfaction. Front Psychol. 2018 Apr 4;9:443. doi: 10.3389/fpsyg.2018.00443. eCollection 2018. PMID 29670559
- [Background] Kasaeian A, Weidenauer C, Hautzinger M, Randler C. Reproductive Success, Relationship Orientation, and Sexual Behavior in Heterosexuals: Relationship With Chronotype, Sleep, and Sex. Evol Psychol. 2019 Jul-Sep;17(3):1474704919859760. doi: 10.1177/1474704919859760. PMID 31272215